CLINICAL TRIAL: NCT01357304
Title: Randomized Controlled Trial of Group Treatment With Physical Activity Referral in a Primary Health Care Setting
Brief Title: 10 Prescriptions an Hour. Group Treatment and Physical Activity Referral in a Primary Health Care Setting
Acronym: 10PAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2011/95
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes; Hypertension
Keywords: Group treatment; Physical activity referral; Type 2 diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group treatment and PAR (Experimental)
  Interventions: Behavioral: Group treatment and PAR
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Group treatment and PAR — Group treatment (8-12 patients per group) involving an empowerment-based process and the 5-A model and including PAR. Two group sessions, 6 months apart. The estimated total time for both group sessions together is 100 minutes.
  Arms: Group treatment and PAR

SUMMARY:
The purpose of this study is to determine the effects of group treatment including physical activity referral (PAR) on level of physical activity and quality of life in patients diagnosed with type 2 diabetes and/or hypertension in a primary health care setting

DETAILED DESCRIPTION:
A sedentary lifestyle and low levels of physical activity in populations are major health problems today and contribute substantially to poor health and diseases such as type 2 diabetes and hypertension. An increased and systematic effort to increase physical activity in the Swedish population in general, and in patients with type 2 diabetes/hypertension in particular, is important. Written prescriptions of physical activity with follow-up (i.e., PAR), is a cost-efficient way to increase physical activity in individuals.

The aim of this trial is to study whether physical activity is increased by a group method involving PARs in patients with hypertension and/or type 2 diabetes compared with a control group that receives usual care in the same primary care setting. Follow-up will be performed at 6 and 12 months.

This trial is being conducted to determine whether it is possible to offer PARs to more patients in a way that requires less effort and resources. The intervention in this study requires 10 minutes of a health care worker's time per patient during a 6-month period. Each patient requires 100 minutes with an instructor who oversees the group intervention.

Group treatment is given 3 weeks after baseline and at 6 months. Follow-up at 12 months involves data collection, but no intervention.

An empowerment process, with the 5-A-model as framework, will be used in the clinical intervention.

All participants will be required to fill in questionnaires and wear an ActiGraph GTM1/GTM3 for 7 days at baseline and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension or type 2 diabetes since 10-09-2009 at St Hans Primary Health Care Center, Lund, Sweden

Exclusion criteria:

* Dementia
* Psychosis
* Drug abuse
* Mental retardation
* Inability to walk without assistance
* Inability to speak Swedish

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Physical activity level | Up to 1 year
  Physical activity level is measured with an Actigraph GTM1/3. Overall physical activity, and total accumulated time and bouts of time in different categories of physical activity, will be determined according to count thresholds. Additonally subjective measurements of physical acidity are made using a questionnaire were questions about self-reported physical activity are reported (the International Physical Activity Questionnaire; IPAQ). Subjectively measured physical activity will be expressed as MET-minutes/week.

SECONDARY OUTCOMES:
Quality of life, measured using the EQ-5D questionnaire | 1 year
  EQ-5D, a validated instrument that classifies health according to five items (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each of which has three alternatives ("no problem", "moderate problem" and "severe problem"). Combining the answers gives an index with a score of between 0.59 and 1.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Primary Health Care Research, Lund University/Region Skane, Malmo, Sweden